CLINICAL TRIAL: NCT01028950
Title: A Multi-center, Open Label Study With YM150, a Direct Factor Xa Inhibitor for Prevention of Venous Thromboembolism in Patients With Acute Medical Illness
Brief Title: YM150 for Prevention of Venous Thromboembolism in Patients With Acute Medical Illness
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Director, Astellas Pharma, Inc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 150-CL-044
Record Dates: First submitted 2009-12-07; First posted 2009-12-09 (Estimated); Last update posted 2010-06-16 (Estimated); Status verified 2010-06

CONDITIONS: Venous Thromboembolism
Keywords: YM150; Bleeding; VTE; FXa inhibitor; Deep Vein Thrombosis; Venous thromboembolism
MeSH Terms: conditions — Venous Thromboembolism; Hemorrhage; Venous Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- YM150 group (Experimental)
  Interventions: Drug: YM150

INTERVENTIONS:
Drug: YM150 — oral

SUMMARY:
To evaluate the safety and efficacy of the oral dose of YM150 for prevention of venous thromboembolism (VTE) in patients with acute medical illness.

ELIGIBILITY:
Inclusion Criteria:

* Patient is hospitalized within 2 days before the study and has more than 1 basic VTE risks
* Complete bed rest is required in the fist day of hospitalization and at least 4 days hospitalization
* Written informed consent obtained

Exclusion Criteria:

* Subject has history of deep vein thrombosis and/or pulmonary embolism
* Subject has a hemorrhagic disorder and/or coagulation disorder
* Subject has had clinically important bleeding occurred within 90 days prior to obtaining informed consent
* Subject has an acute bacterial endocarditis
* Subject has uncontrolled severe or moderate hypertension, retinopathy, myocardial infarction or stroke
* Subject is receiving anticoagulants/antiplatelet agents
* Subject has a body weight less than 40 kg
* Major trauma, major surgery, eye, spinal cord and/or brain surgery within 90 days prior to obtaining informed consent, or the subject scheduled for these surgeries during the study periods

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2009-05; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Composite assessment of VTE events and all cause death | Until day 28

SECONDARY OUTCOMES:
Incidence of bleeding events | Until day 28

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (5):
- Japan (5):
  - Chugoku
  - Chūbu
  - Kansai
  - Kantou
  - Tōhoku